CLINICAL TRIAL: NCT04766307
Title: A Randomized Multicenter Clinical Trial of a New Treatment for Primary Smear- Positive Pulmonary Tuberculosis With Interleukin-2
Brief Title: A New Treatment for Primary Smear-positive Pulmonary Tuberculosis With Interleukin-2
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Chest Hospital (Other)
Responsible Party: Principal Investigator, Chu naihu, Director,TB Department, Beijing Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015ZX10003001-002
Record Dates: First submitted 2017-12-20; First posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Tuberculosis, Pulmonary
Keywords: pulmonary tuberculosis; interleukin-2; clinical trial
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- experimental group (Experimental): Experimental group regimen:2H(Isoniazid)R(Rifampicin)Z(Pyrazinamide)E(Ethambutol)/4HR+Interleukin-2 （500000 units daily, subcutaneous injection in the first month）
  Dosage: isoniazid 300mg(given once daily),rifampin 450mg(less than 50kg,given once daily) or 600mg(more than 50kg,given once daily),pyrazinamide 1500mg(less than 50kg,given once daily) or 30mg/kg(more than 50kg,given once daily),ethambutol 750mg(less than 50kg,given once daily) or 1000mg(more than 50kg,given once daily).
  Interventions: Drug: Interleukin-2
- Control regimen group (Active Comparator): The control group regimen: 2H(Isoniazid)R(Rifampicin)Z(Pyrazinamide)E(Ethambutol)/4HR
  Dosage: isoniazid 300mg(given once daily),rifampin 450mg(less than 50kg,given once daily) or 600mg(more than 50kg,given once daily),pyrazinamide 1500mg(less than 50kg,given once daily) or 30mg/kg(more than 50kg,given once daily),ethambutol 750mg(less than 50kg,given once daily) or 1000mg(more than 50kg,given once daily).
  Interventions: Drug: Interleukin-2

INTERVENTIONS:
Drug: Interleukin-2 — Interleukin 2 (IL-2) is a pleiotropic cytokine that is produced after antigen activation and plays crucial roles in the immune response. IL-2 secreted by activated T cells is central to the development of an immune response to infection, promoting the differentiation and proliferation of lymphoid cells. This hydrophobic molecule and the various cytokines that it elicits regulates the behavior of T and B lymphocytes, monocytes/macrophages, natural killer (NK) cells, and neutrophils. IL-2 therapy regimens are expected to limit mycobacterial replication. Early clinical trials with IL-2 demonstrated that IL-2 immunotherapy may be useful in controlling infectious disease.
  Other Names: IL-2

SUMMARY:
The purpose of the study is to compare the efficacy and safety of standard chemotherapy regimen 2HRZE/4HR plus IL-2 and standard regimen 2HRZE/4HR for newly diagnosed smear positive pulmonary tuberculosis.

DETAILED DESCRIPTION:
1. Design:The study is a multi-center, randomized, controlled, open clinical trial.
2. Population:Initial smear positive pulmonary tuberculosis patients who fulfill the inclusion and exclusion criteria.
3. Investigational regimens:

   Experimental group regimen:2HRZE/4HR+Interleukin-2 （500000 units daily, subcutaneous injection in the first month） The control group regimen: 2HRZE/4HR Dosage: isoniazid 300mg(given once daily),rifampin 450mg(less than 50kg,given once daily) or 600mg(more than 50kg,given once daily),pyrazinamide 1500mg(less than 50kg,given once daily) or 30mg/kg(more than 50kg,given once daily),ethambutol 750mg(less than 50kg,given once daily) or 1000mg(more than 50kg,given once daily).
4. Primary and Secondary outcome measures:

primary efficacy outcome measures:(a)Negative conversion rate of sputum bacteria. (b)Sputum smear conversion proportion at the treatment completion .

secondary efficacy outcome measure:Recurrence rate after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Is willing and able to give informed consent to participate in the trial treatment and follow-up (signed or witnessed consent if the patient is illiterate).
2. Is aged 18-65 years.
3. Chest X-ray showed that there were active tuberculosis foci in the lungs with one of the following cases: (1) sputum specimens (or sputum and bronchial lavage fluid) were 2+ once or 1+ twice ; (2) sputum smear positive and sputum X-pert positive.
4. Newly diagnosed cases receiving anti-TB treatment for less than one month.
5. No other immune preparations （such as: thymosin，IFN-y，BCG-PSN，Mycobacterium vaccae，Utilins，lentinan ）were used in the past 3 months.
6. the urine analysis of Women of childbearing age are negative and agree to use the efficient contraception during the study period.

Exclusion Criteria:

1. Has a known allergy to any drug of treatment regimens.
2. There are serious complications or impaired renal function (serum creatinine is 1.5 times higher than the normal limit) or impaired liver function (ALT or AST levels are 3 times higher than the normal limit); hemoglobin is less than 7.0g/dl. Platelets less than 50x109/L.
3. Complication with Diabetic.
4. The screening diagnosis was isoniazid resistance or rifampin resistance
5. There are serious cardiovascular diseases, such as heart failure, hypertension, arrhythmia or post myocardial infarction state.
6. Is known to be pregnant or breast-feeding.
7. Karnofsky score is less than 50%.
8. Is taking any clinical trial in the past 3 months.
9. Is critically ill, and in the judgment of the investigator, not fit for the study or unlikely to complete the full course of study.
10. HIV is positive or AIDS patients.
11. Has Non tuberculous mycobacterial lung disease.
12. Merge with extra pulmonary tuberculosis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2016-07-20 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary study endpoint was the proportion of subjects who had converted their sputum cultures to negative at the end of treatment. | two-month course intensive phase treatment, followed by a four-month consolidation phase treatment.Some TB patients with cavity should receive 9 total months (7 months of continuation therapy after the initial 2-month intensive phase).
  A cure was defined as who was smear- or culture-negative in the last month of treatment and on at least one previous occasion. Treatment completion was defined as patients who completed treatment but who does not have a negative sputum smear or culture result in the last month of treatment and on at least one previous occasion. Treatment failure was defined as patients whose sputum smear or culture is positive at 5 months or later during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Naihui Chu, PhD, Principal Investigator — Beijing Chest Hospital
Locations (16):
- China (16):
  - the Second hospital of Fuyang, Fuyang, Anhui
  - Fuzhou Chest Hospital, Fuzhou, Fujian
  - Shenzhen third people's Hospital, Shenzhen, Guangzhou
  - Guiyang Public Health Treatment Center, Guiyang, Guizhou
  - The Infectious Hospital of Handan, Handan, Hebei
  - Hebei Chest Hospital, Shijiazhuang, Hebei
  - Jiamusi Insititute For Tuberculosis Control, Jiamusi, Heilongjiang
  - The Infectious Hospital of mudanjiang, Mudanjiang, Heilongjiang
  - Zhengzhou Sixth People's Hospital, Zhengzhou, Henan
  - the central hospital of Changsha, Changsha, Hunan
  - the people's hospital of Jiangsu province, Nanjing, Jiangsu
  - Jiangxi Chest Hospital, Nanchang, Jiangxi
  - Dalian Tuberculosis Hospital, Dalian, Liaoning
  - Qingdao Chest Hospital, Qingdao, Shandong
  - Taiyuan Fourth People's Hospital, Taiyuan, Shanxi
  - Xian Chest Hospital, Xi’an, Shanxi